CLINICAL TRIAL: NCT05467644
Title: Treatment of Fracture Related Infection in Latin America. International Multicenter Study
Brief Title: Treatment of Fracture Related Infection in Latin America.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Manoel Victorino Hospital (Other Government)
Collaborators: AO Trauma Latin America (Unknown); Centro Médico Nacional de Occidente IMSS (Unknown); University of Campinas, Brazil (Other); Hospital Municipal Miguel Couto (Other); Hospital Italiano de Buenos Aires (Other); Hospital Pablo Tobón Uribe (Other)
Responsible Party: Principal Investigator, Matheus Lemos Azi, Principal Investigator, Manoel Victorino Hospital
Other Study IDs: FRI LATIN AMERICA - AOLAT
Record Dates: First submitted 2022-07-06; First posted 2022-07-20 (Actual); Last update posted 2022-07-20 (Actual); Status verified 2022-07

CONDITIONS: Fracture; Osteomyelitis; Soft Tissue Injuries; Bone Loss
Keywords: Fracture; Osteomyelitis; Soft Tissue Injuries; Bone Loss
MeSH Terms: conditions — Fractures, Bone; Osteomyelitis; Soft Tissue Injuries; Bone Diseases, Metabolic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Treatment of Fracture Related Infection — Observational Retrospective Study. Only one group. Patients diagnosed with fracture-related infection and submitted to surgical treatment

SUMMARY:
Postoperative bone infection is a severe complication in the treatment of fractures and is more frequent than in elective joint replacement surgeries. Surgical treatment is based on meticulous debridement of bone and soft tissue, dead space management, soft tissue reconstruction when necessary, and restoration of bony stability in the non-union fracture. In addition, local antibiotic therapy is recommended in certain circumstances. This study aims to evaluate the results of surgical treatment of fracture-related infection in Latin America.

DETAILED DESCRIPTION:
Research question: What are the characteristics and the diagnostic and therapeutic approach of patients with fracture-related infections (FRI) managed in various centers in Latin America?

Objectives:

General objective Describe the treatment of FRI in different institutions in Latin America, emphasizing the diagnostic process and the surgical and medical approach to this type of patient.

Specific objectives:

To analyze the usefulness of the criteria proposed by the expert consensus for diagnosing FRI.

Describe surgical treatment strategies in patients with FRI. Describe the microbiological profile of FRI in Latin American centers To explore variables associated with outcomes. Describe strategies for managing soft tissue defects associated with FRI. Describe the results regarding patients' quality of life with FRI.

Methodology:

Type of study: Observational retrospective cohort study

Outcomes to evaluate:

Infectious relapse: Presence of confirmatory or suggestive clinical signs of infection related to fractures, according to the FRI consensus criteria, within the first year of follow-up after the main surgery for the treatment of infection, and that motivates an intervention additional (Surgery or additional antibiotics) Consolidation: defined as clinical and radiological consolidation. Clinical consolidation - the absence of pain on local palpation and with load or walking. Radiological consolidation - Presence of bone trabeculae in the fracture line in the four cortices of the two standard radiological projections.

Complications: Defined as any adverse event that requires surgery for treatment. It can be "immediate" (those requiring an additional surgical procedure within up to 30 days of treatment of the infection. Examples: hematoma, debridement, change of fixators, change of implant, even if partial) or "late" ( those that required surgical procedure after 30 days of definitive treatment (for example debridement, implant failure, bone grafting).

Proposed statistical analysis: Descriptive statistics tools will be used for qualitative variables, absolute and relative frequencies, quantitative variables, measures of central tendency such as mean or median, and measures of dispersion such as standard deviation or interquartile range, according to the distribution of the variables. Univariate analyses will be performed to explore the relationship of different variables with the risk of infectious relapse, treatment failure, and amputation. All statistical analyzes will be executed in SPSS Statistics® v20 (IBM, Chicago, IL).

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (18 years or older)
* Infection after surgical fracture treatment occurred 90 days after the initial surgery.
* Definitive treatment in one of the centers involved
* Hospital admission from January 1, 2018, to December 31, 2020
* Minimum outpatient follow-up period of one year after the main surgery to treat the infection, assess the quality of life, and control of the infection.

Exclusion Criteria:

* Incomplete medical records

Min Age: 16 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Patients diagnosed with Fracture-related Infection
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2022-09-01 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Usefulness of the FRI diagnosing criteria | at least 6 months after infection treatment
  To analyze the usefulness of the criteria proposed by the expert consensus for diagnosing fractures-related infections.

SECONDARY OUTCOMES:
Surgical treatment | at least 12 months after infection treatment
  Describe the strategies of surgical treatment in patients with infections related to fractures
Microbiological profile | just after infection treatment
  Describe the microbiological profile of fracture-related infections in Latin American centers.
Variables associated with outcomes | at least 12 months after infection treatment
  To explore variables associated with the outcome of fracture-related infection control
Strategies for the management of soft tissue defects | at least 6 months after infection treatment
  Describe the strategies for the management of soft tissue defects associated with infections related to fractures.
Quality of life - EQ-5D-3L | at least 12 months after infection treatment
  Describe the results in terms of the quality of life of patients with infections related to fractures

CONTACTS AND LOCATIONS:
Locations (1):
- Manoel Victorino Hospital, Salvador, Estado de Bahia, Brazil

IPD SHARING:
Plan to Share IPD: Undecided
Six countries are involved in the study, and they have different regulations regarding handling patient data. Therefore, researchers will assess data sharing during the data analysis phase of the study.

REFERENCES:
- [Background] Walter G, Kemmerer M, Kappler C, Hoffmann R. Treatment algorithms for chronic osteomyelitis. Dtsch Arztebl Int. 2012 Apr;109(14):257-64. doi: 10.3238/arztebl.2012.0257. Epub 2012 Apr 6. PMID 22536302
- [Background] Trampuz A, Zimmerli W. Diagnosis and treatment of infections associated with fracture-fixation devices. Injury. 2006 May;37 Suppl 2:S59-66. doi: 10.1016/j.injury.2006.04.010. PMID 16651073
- [Background] Steinmetz S, Wernly D, Moerenhout K, Trampuz A, Borens O. Infection after fracture fixation. EFORT Open Rev. 2019 Jul 15;4(7):468-475. doi: 10.1302/2058-5241.4.180093. eCollection 2019 Jul. PMID 31423330
- [Background] Alcantara JE JUNIOR, Aguiar RA, Sampaio JGL NETO, Azi ML, Sadigursky D, Alencar DF. FACTORS ASSOCIATED WITH THE DEVELOPMENT OF EARLY INFECTION AFTER SURGICAL TREATMENT OF FRACTURES. Acta Ortop Bras. 2018 Jan-Feb;26(1):22-26. doi: 10.1590/1413-785220182601173883. PMID 29977139
- [Background] Metsemakers WJ, Morgenstern M, McNally MA, Moriarty TF, McFadyen I, Scarborough M, Athanasou NA, Ochsner PE, Kuehl R, Raschke M, Borens O, Xie Z, Velkes S, Hungerer S, Kates SL, Zalavras C, Giannoudis PV, Richards RG, Verhofstad MHJ. Fracture-related infection: A consensus on definition from an international expert group. Injury. 2018 Mar;49(3):505-510. doi: 10.1016/j.injury.2017.08.040. Epub 2017 Aug 24. PMID 28867644
- [Background] Depypere M, Morgenstern M, Kuehl R, Senneville E, Moriarty TF, Obremskey WT, Zimmerli W, Trampuz A, Lagrou K, Metsemakers WJ. Pathogenesis and management of fracture-related infection. Clin Microbiol Infect. 2020 May;26(5):572-578. doi: 10.1016/j.cmi.2019.08.006. Epub 2019 Aug 22. PMID 31446152
- [Background] Zimmerli W, Sendi P. Orthopaedic biofilm infections. APMIS. 2017 Apr;125(4):353-364. doi: 10.1111/apm.12687. PMID 28407423
- [Background] Hotchen AJ, McNally MA, Sendi P. The Classification of Long Bone Osteomyelitis: A Systemic Review of the Literature. J Bone Jt Infect. 2017 Sep 12;2(4):167-174. doi: 10.7150/jbji.21050. eCollection 2017. PMID 29119075
- [Background] Morgenstern M, Moriarty TF, Kuehl R, Richards RG, McNally MA, Verhofstad MHJ, Borens O, Zalavras C, Raschke M, Kates SL, Metsemakers WJ. International survey among orthopaedic trauma surgeons: Lack of a definition of fracture-related infection. Injury. 2018 Mar;49(3):491-496. doi: 10.1016/j.injury.2018.02.001. Epub 2018 Feb 6. PMID 29433799
- [Background] Metsemakers WJ, Kuehl R, Moriarty TF, Richards RG, Verhofstad MHJ, Borens O, Kates S, Morgenstern M. Infection after fracture fixation: Current surgical and microbiological concepts. Injury. 2018 Mar;49(3):511-522. doi: 10.1016/j.injury.2016.09.019. Epub 2016 Sep 11. PMID 27639601
- [Background] Bezstarosti H, Van Lieshout EMM, Voskamp LW, Kortram K, Obremskey W, McNally MA, Metsemakers WJ, Verhofstad MHJ. Insights into treatment and outcome of fracture-related infection: a systematic literature review. Arch Orthop Trauma Surg. 2019 Jan;139(1):61-72. doi: 10.1007/s00402-018-3048-0. Epub 2018 Oct 20. PMID 30343322
- [Background] Govaert GAM, Kuehl R, Atkins BL, Trampuz A, Morgenstern M, Obremskey WT, Verhofstad MHJ, McNally MA, Metsemakers WJ; Fracture-Related Infection (FRI) Consensus Group. Diagnosing Fracture-Related Infection: Current Concepts and Recommendations. J Orthop Trauma. 2020 Jan;34(1):8-17. doi: 10.1097/BOT.0000000000001614. PMID 31855973
- [Background] Metsemakers WJ, Fragomen AT, Moriarty TF, Morgenstern M, Egol KA, Zalavras C, Obremskey WT, Raschke M, McNally MA; Fracture-Related Infection (FRI) consensus group. Evidence-Based Recommendations for Local Antimicrobial Strategies and Dead Space Management in Fracture-Related Infection. J Orthop Trauma. 2020 Jan;34(1):18-29. doi: 10.1097/BOT.0000000000001615. PMID 31464858

DOCUMENTS (1):
  • Study Protocol (2021-07-01): https://cdn.clinicaltrials.gov/large-docs/44/NCT05467644/Prot_000.pdf